CLINICAL TRIAL: NCT02276898
Title: A Randomized-Controlled Trial of Inhaled Hypertonic Saline (7%) to Evaluate the Lung Clearance Index as a Short-term Pharmacodynamic Biomarker in Patients With Cystic Fibrosis.
Brief Title: A Randomized-Controlled Trial of Inhaled Hypertonic Saline (7%) to Evaluate the Lung Clearance Index
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Reshma Amin, Staff Respirologist, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1000024909
Record Dates: First submitted 2014-10-22; First posted 2014-10-28 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Cystic Fibrosis
Keywords: pediatric; lung clearance index; Multiple Breath Washout; Hypertonic Saline
MeSH Terms: conditions — Cystic Fibrosis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypertonic Saline (Active Comparator): The treatment intervention is 1 inhalation of 7% hypertonic saline (4ml)
  Interventions: Drug: Hypertonic Saline 7%
- Isotonic Saline (Placebo Comparator): The placebo intervention is 1 inhalation of 0.9% isotonic saline
  Interventions: Drug: Isotonic Saline 0.9% (Placebo)

INTERVENTIONS:
Drug: Hypertonic Saline 7% — PARI Hyper-Sal™ Sodium Chloride Solution - 7%
  Arms: Hypertonic Saline
Drug: Isotonic Saline 0.9% (Placebo)
  Arms: Isotonic Saline

SUMMARY:
The Lung Clearance Index (LCI) is a non invasive measure of lung function that is more sensitive than FEV1. It can be used to measure lung function in children younger than 6 years of age. Therefore, it has a future role in assessing novel therapeutics in the Cystic Fibrosis (CF) population. As such, determining if it can be used as a short term pharmacodynamic biomarker is paramount.

DETAILED DESCRIPTION:
Inhaled Hypertonic saline (7%) is a treatment intervention for Cystic Fibrosis patients and has previously been shown to improve lung function and decrease the number of pulmonary exacerbations. The Cystic Fibrosis Transmembrane Regulator Gene (CFTR) protein is essential for maintaining fluid and electrolyte homeostasis in the lung and CFTR defects cause depletion of the periciliary liquid layer which results in impaired mucociliary clearance. Inhaled hypertonic saline (7%) acts as an osmotic agent in the lungs; it repletes the airway surface liquid (ASL) and improves mucociliary clearance.

In addition, we have recently demonstrated that the Lung Clearance Index (LCI) is also a responsive outcome measure. In an intervention study in which patients were treated with hypertonic saline inhalation twice daily for 28 days, LCI but not FEV1 significantly improved in 17 pediatric Cystic Fibrosis (CF) patients with mild lung disease. In this study, LCI was more sensitive to a change in response to treatment than spirometry in a small number of patients. However, it still remains unknown if the LCI will be able to detect a treatment effect on a shorter time scale after an intervention. Its use as a short-term pharmacodynamic biomarker in CF patients remains unknown. The ability of the LCI to detect treatment effects within hours after an intervention would be invaluable to the development of new therapeutic interventions for CF patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF as defined by two or more clinical features of CF and a documented sweat chloride > 60 mEq/L by quantitative pilocarpine iontophoresis test or a genotype showing two well characterized disease causing mutations
* Informed consent and verbal assent (as appropriate) provided by the subject's parent or legal guardian and the subject
* At least six years of age at enrolment
* Able to perform reproducible spirometry meeting American Thoracic Society standards
* Pre-bronchodilator FEV1 % predicted > or equal to 40 % predicted
* Ability to perform a reproducible LCI maneuver at screening

Exclusion Criteria:

* Known respiratory culture positive for Burkholderia cepacia
* Previous lung transplantation
* Use of intravenous antibiotics within 14 days of screening
* Use of oral antibiotics including prophylactic antibiotics (e.g., augmentin, tetracycline, cloxacillin, cephalosporins, septra, bactrim) within 14 days of screening
* Initiation of a new maintenance (e.g high dose ibuprofen, Pulmozyme®, aerosolized antibiotics) within 14 days of screening
* Use of systemic corticosteroids within 14 days of screening
* Investigational drug use within 30 days of screening
* Use of hypertonic saline (7%) < 4 weeks before screening or outside of the study protocol
* Participation in any therapeutic clinical study <4 weeks or, 5 half-lives, whichever is longer, before screening
* Smoking < 3 months before screening
* Presence of a condition or abnormality that in the opinion of the site investigator would compromise the safety of the subject or the quality of the data

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Lung Clearance Index | Baseline to 24 hrs post dose
  The change in the Lung Clearance Index as measured by nitrogen washout between baseline and 24 hours after each inhalation of Hypertonic Saline (7%) and Isotonic Saline (0.9%)

SECONDARY OUTCOMES:
Pulmonary Function Testing | Baseline, 1,2,4 and 24hrs post-dose
  Forced Expiratory Volume in one second (FEV1) % predicted, Forced Expiratory Vital Capacity (FVC) % predicted and Forced Expiratory Flow rate (FEF) 25-75 % predicted will be measured using spirometry.
Lung Clearance Index measured using Mass Spectroscopy | Baseline, 1,2,4 and 24 hrs post dose
  The multiple breath washout will be performed in the classical method using a mass spectroscopy (MS): each test consists of two phases: a wash-in phase and washout phase using an inert dry gas mixture containing 4% Sulfur hexafluoride (SF6), 4% He, 21% oxygen and balance nitrogen.
Lung Clearance Index measured using Nitrogen Washout | Baseline, 1,2, 4hrs post dose
  The change in the Lung Clearance Index as measured by nitrogen washout between baseline and 1,2 and 4 hours after each inhalation of Hypertonic Saline (7%) and Isotonic Saline (0.9%)

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Amin, MD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - St. Michaels Hospital, Toronto, Ontario